CLINICAL TRIAL: NCT05702736
Title: The Effect of Logotherapy-Based Intervention on Depression Patients on Depression, Psychological Pain, and Meaning of Life: Follow-Up Study With Control Group
Brief Title: The Effect of Logotherapy-Based Intervention on Depression Patients on Depression,Psychological Pain and Meaning of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Merve Uğuryol Ünal, Research Assistant, Phd Student, Ege University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-3T/42; 20-3T/42 (Other: Ege University Medical Research Ethics Committee)
Record Dates: First submitted 2023-01-08; First posted 2023-01-27 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Beck Depression Inventory, Psychache Scale, Meaning of Life Questionnaire was applied to intervention group as a pre-test. Inaddition to the Standard treatment, the intervention group received a logotherapy-based intervention. Beck Depression Inventory, Psychache Scale, Meaning of Life Questionnaire was applied to intervention group as a post test and follow up test.
  Interventions: Behavioral: logotherapy-based intervention
- Control group (No Intervention): Beck Depression Inventory, Psychache Scale, Meaning of Life Questionnaire was applied to control group as a pre-test. The control group received only standard treatment. Beck Depression Inventory, Psychache Scale, Meaning of Life Questionnaire was applied to control group as a post test and follow up test.

INTERVENTIONS:
Behavioral: logotherapy-based intervention — Logotherapy-based intervention was administered to the individuals in the intervention group as a total of eight sessions, once a week.
  Arms: Intervention group

SUMMARY:
The goal of this interventional study is to compare in logotherapy-based intervention practiced to depressed patients on depression, psychological pain and meaning of life. The main questions it aims to answer are:

* Is the logotherapy-based intervention practiced in addition to the standard treatment in depression patients effective in reducing the depression levels of the patients?
* Is the logotherapy-based intervention practiced in addition to the standard treatment in depression patients effective in reducing the psychological pain levels of the patients?
* Is the logotherapy-based intervention practiced in addition to the standard treatment in depression patients effective in increasing the patients' level of meaning to life? Participants will be done online interview once a week for eight sessions. Researchers will compare intervention and control groups to see if logotherapy-based intervention practiced effect depression, psychological pain and meaning of life levels.

DETAILED DESCRIPTION:
The research was conducted to examine the effect of logotherapy-based intervention practiced to depressed patients on depression, psychological pain and meaning of life.

The research is in a quasi-experimental research design with pre-test post-test follow-up measurement, control group. Sample selection was carried out in two stages, and in the first stage, 48 patients diagnosed with depression between September 2020 and September 2022 were referred to the researcher by the polyclinic physician. The patients were evaluated within the scope of the inclusion criteria of the study, and 32 patients with a diagnosis of depression, aged 18-65 years, voluntarily aged between 18-65, who scored 17 points or more from the Beck Depression Inventory, were accepted into the study. Patients were assigned to intervention and control groups, respectively. A total of 28 patients, 12 intervention and 16 control groups, completed the study. "Descriptive Information Form", "Beck Depression Inventory", "Psychache Scale" and "Meaning of Life Questionnaire" were used as data collection tools in the study. Online logotherapy-based intervention was administered to the individuals in the intervention group as a total of eight sessions, once a week. In order to evaluate the effect of logotherapy-based intervention, Beck Depression Inventory, Psychache Scaleand Meaning of Life Questionnaire were administered to all individuals in the sample group at time series points (pretest, posttest, follow-up test at 3rd month). In the analysis of the data, descriptive statistics, independent t-test, chi-square analysis, analysis of variance in repeated measurements, Bonferroni correction were applied.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-65
* Having been diagnosed with depression
* A score of 17 or higher on the Beck Depression Inventory
* Willingness and willingness to participate in the research
* Completed at least six interviews

Exclusion Criteria:

* Having an active risk of suicide
* Having psychotic symptoms
* Having a psychiatric comorbidity
* Using antipsychotic medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2022-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esra ENGİN, Study Chair — Ege University
Locations (1):
- Ege University Faculty of Nursing, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 16 | 16
Completed | 12 | 16
Not Completed | 4 | 0
Not completed — 2 patients didn't participate in the study voluntarily. | 2 | 0
Not completed — 2 patients didn't complete 6 interviews. | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 12 | 16 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 16 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Data were collected with a descriptive information form.
  years | 36.25 (10.72) | 34.94 (10.69) | 35.50 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 3 | 6 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 12 | 16 | 28
Beck Depression Inventory Pretest [Mean (Standard Deviation); unit: scores on a scale] — Beck Depression Inventory (BDI) The inventory measures depression level.The inventory assesses physical, emotional, cognitive and motivational components. The four-point Likert-type scale comprises of 21 questions. The scale has a minimum score of 0 and a maximum score of 63. As the total score increases, the depression level also increases. The scale score graded depression into four levels: normal (0-9 points), mild (10-16 points), moderate (17-29 points) and severe (30-63 points)
  scores on a scale | 33.25 (9.41) | 29.62 (8.49) | 31.18 (8.92)
Psychache Scale [Mean (Standard Deviation); unit: scores on a scale] — Psychache Scale was developed to assess psychological pain. The five-point Likert-type scale consists of 13 questions. The scale has a minimum score of 13 and a maximum score of 65. As the total score increases, the psychache level increases. Decreased "Psychache Scale" scores of the intervention group in post test and follow-up measurements after logotherapy-based intervention.
  scores on a scale | 50.17 (8.37) | 43.94 (14.00) | 46.61 (12.14)
Meaning in Life Questionnaire [Mean (Standard Deviation); unit: scores on a scale] — Meaning of Life Questionnaire measures the level of meaning that individuals give to life.This seven-point Likert-type scale consists of 10 questions.The scale has a minimum score of 10 and a maximum score of 70. The scale has two subscales. These subscales include the existing meaning in life (5 questions) and the search for meaning in life (5 questions).The total score is obtained by summing the subscale scores. As the total score of the scale increases, individuals' level of meaning in life increases.
  scores on a scale | 35.50 (16.19) | 40.62 (7.05) | 38.43 (11.88)

OUTCOME MEASURES:

1. Primary Outcome: "Beck Depression Inventory" Scores
Description: Beck Depression Inventory (BDI) The inventory measures depression level.The inventory assesses physical, emotional, cognitive and motivational components. The four-point Likert-type scale comprises of 21 questions. The scale has a minimum score of 0 and a maximum score of 63. As the total score increases, the depression level also increases. The scale score graded depression into four levels: normal (0-9 points), mild (10-16 points), moderate (17-29 points) and severe (30-63 points).
Time Frame: post-test (after 8 weeks) and follow-up test (after 3 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention Group: Beck Depression Inventory was applied to intervention group as a pre-test. Inaddition to the Standard treatment, the intervention group received a logotherapy-based intervention. Beck Depression Inventory was applied to intervention group as a post test and follow up test.
  logotherapy-based intervention: Logotherapy-based intervention was administered to the individuals in the intervention group as a total of eight sessions, once a week.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 12 | 16
score on a scale
  Beck Depression Inventory Post Test | 17.75 (9.18) | 30.62 (8.76)
  Beck Depression Inventory Follow Up Test | 13.58 (10.76) | 31.18 (10.44)

2. Primary Outcome: "Psychache Scale" Scores
Description: Psychache Scale was developed to assess psychological pain. The five-point Likert-type scale consists of 13 questions. The scale has a minimum score of 13 and a maximum score of 65. As the total score increases, the psychache level increases.
Time Frame: post-test (after 8 weeks) and follow-up test (after 3 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention Group: Psychache Scale was applied to intervention group as a pre-test. Inaddition to the Standard treatment, the intervention group received a logotherapy-based intervention. Psychache Scale was applied to intervention group as a post test and follow up test.
  logotherapy-based intervention: Logotherapy-based intervention was administered to the individuals in the intervention group as a total of eight sessions, once a week.
- Control Group: Psychache Scale applied to intervention group as a pre-test. Inaddition to the Standard treatment, the intervention group received a logotherapy-based intervention. Psychache Scale was applied to intervention group as a post test and follow up test.
  logotherapy-based intervention: Logotherapy-based intervention was administered to the individuals in the intervention group as a total of eight sessions, once a week.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 12 | 16
score on a scale
  Psychache Scale Post Test | 27.83 (5.90) | 45.81 (13.69)
  Psychache Scale Follow Up Test | 27.83 (11.70) | 46.25 (13.09)

3. Primary Outcome: "Meaning of Life Questionnaire" Scores
Description: Meaning of Life Questionnaire measures the level of meaning that individuals give to life.This seven-point Likert-type scale consists of 10 questions.The scale has a minimum score of 10 and a maximum score of 70. The scale has two subscales. These subscales include the existing meaning in life (5 questions) and the search for meaning in life (5 questions).The total score is obtained by summing the subscale scores. As the total score of the scale increases, individuals' level of meaning in life increases.
Time Frame: post-test (after 8 weeks) and follow-up test (after 3 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Intervention Group: Meaning of Life Questionnaire was applied to intervention group as a pre-test. Inaddition to the Standard treatment, the intervention group received a logotherapy-based intervention. Meaning of Life Questionnaire was applied to intervention group as a post test and follow up test.
  logotherapy-based intervention: Logotherapy-based intervention was administered to the individuals in the intervention group as a total of eight sessions, once a week.
- Control Group: Meaning of Life Questionnaire was applied to control group as a pre-test. The control group received only standard treatment. Meaning of Life Questionnaire was applied to control group as a post test and follow up test.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 12 | 16
score on a scale
  Meaning of Life Questionnaire Post Test | 42.83 (10.89) | 39.25 (6.32)
  Meaning of Life Questionnaire Follow up test | 50.25 (7.17) | 37.81 (6.01)

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this study.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
It is among the limitations that the patients in the intervention and control groups can experience improvement thanks to the use of psychiatric drugs other than logotherapy-based applications. The research was conducted during the Covid-19 pandemic. Face-to-face meetings were held online. Again, depression levels may have been affected since patients had to be forced to stay at home. These possibilities are among the limitations of the research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT05702736/Prot_000.pdf